CLINICAL TRIAL: NCT01915173
Title: Response to Supplement and Placebo in GERD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Gloria Y. Yeh, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012P000409; IND 117358 (Other: FDA)
Record Dates: First submitted 2013-07-30; First posted 2013-08-02 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2016-12

CONDITIONS: Gastroesophageal Reflux Disease (GERD); Heartburn; Dyspepsia
Keywords: Gastroesophageal reflux disease (GERD); Heartburn; Dyspepsia
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn; Dyspepsia | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Supplement + Expanded Interview (Experimental): Supplement, 2 tablets sublingually 3 times a day for 2 weeks.
  Interventions: Drug: Supplement; Behavioral: Expanded Interview
- Placebo + Standard Interview (Placebo Comparator): Placebo, 2 tablets sublingually 3 times a day for 2 weeks.
  Interventions: Drug: Placebo; Behavioral: Standard Interview
- Supplement + Standard Interview (Experimental): Supplement, 2 tablets sublingually 3 times a day for 2 weeks.
  Interventions: Drug: Supplement; Behavioral: Standard Interview
- Placebo + Expanded Interview (Placebo Comparator): Placebo, 2 tablets sublingually 3 times a day for 2 weeks.
  Interventions: Drug: Placebo; Behavioral: Expanded Interview

INTERVENTIONS:
Drug: Supplement — Abies nigra 4C, Carbo vegetabilis 4C, Nux vomica 4C, and Robinia pseudoacacia 4C
  Arms: Supplement + Expanded Interview; Supplement + Standard Interview
Drug: Placebo — Lactose tablets
  Arms: Placebo + Expanded Interview; Placebo + Standard Interview
Behavioral: Expanded Interview
  Arms: Placebo + Expanded Interview; Supplement + Expanded Interview
Behavioral: Standard Interview
  Arms: Placebo + Standard Interview; Supplement + Standard Interview

SUMMARY:
The purpose of this study is to investigate the effects of a widely available over the counter supplement marketed for heartburn symptoms on symptoms and health-related quality of life in patients with gastroesophageal reflux disease (GERD). This study is designed as a pilot trial to assess safety and feasibility and to provide preliminary estimates of effect sizes.

ELIGIBILITY:
Inclusion Criteria:

* Adult humans age 18-80.
* Fluency in written and spoken English.
* Heartburn symptoms 3 or more days per week for the past month.

Exclusion Criteria:

* Individuals taking a proton pump inhibitor (PPI) or H2 receptor blocker with a dose change within 2 weeks of the initial study visit.
* Individuals with Crohns disease, systemic sclerosis, known active ulcer disease, gastric cancer, Barrett's esophagitis
* Significant pain or difficulty with swallowing
* Heavy alcohol use (defined by > 6 drinks/week for women and > 13 drinks/week for men)
* Concurrent pregnancy
* Dementia
* Uncontrolled psychiatric disease
* Individuals unable to complete a paper symptom diary for 6 of 7 days prior to their baseline visit
* Subjects whose symptoms are predominantly dyspeptic more than heartburn or reflux
* Subjects who have used homeopathy for GI symptoms or have received constitutional homeopathic treatment within the past 2 weeks
* Subjects taking herbal products or other supplements for GERD or dyspepsia related symptoms (includes peppermint oil)
* Subjects who have taken > 12 doses of NSAIDS within the prior 30 days (aspirin ≤ 325 mg daily is allowed)
* Subjects with lactose intolerance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Dossett, MD, PhD, MPH, Study Director — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Dossett ML, Mu L, Davis RB, Bell IR, Lembo AJ, Kaptchuk TJ, Yeh GY. Patient-Provider Interactions Affect Symptoms in Gastroesophageal Reflux Disease: A Pilot Randomized, Double-Blind, Placebo-Controlled Trial. PLoS One. 2015 Sep 30;10(9):e0136855. doi: 10.1371/journal.pone.0136855. eCollection 2015. PMID 26422466
- See also: study manuscript — http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0136855

RESULTS

PARTICIPANT FLOW:
Groups:
- Supplement + Expanded Interview: Supplement, 2 tablets sublingually 3 times a day for 2 weeks.
  Supplement = Acidil: Abies nigra 4C, Carbo vegetabilis 4C, Nux vomica 4C, and Robinia pseudoacacia 4C
  Expanded Interview
- Placebo + Standard Interview: Placebo, 2 tablets sublingually 3 times a day for 2 weeks.
  Placebo: Lactose tablets
  Standard Interview
- Supplement + Standard Interview: Supplement, 2 tablets sublingually 3 times a day for 2 weeks.
  Supplement = Acidil: Abies nigra 4C, Carbo vegetabilis 4C, Nux vomica 4C, and Robinia pseudoacacia 4C
  Standard Interview
- Placebo + Expanded Interview: Placebo, 2 tablets sublingually 3 times a day for 2 weeks.
  Placebo: Lactose tablets
  Expanded Interview
Period: Overall Study
Arm/Group | Supplement + Expanded Interview | Placebo + Standard Interview | Supplement + Standard Interview | Placebo + Expanded Interview
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Standard Interview | Supplement + Standard Interview | Placebo + Expanded Interview | Supplement + Expanded Interview | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 5 | 5 | 17
  >=65 years | 3 | 2 | 1 | 1 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (14) | 64 (6.3) | 54 (9.9) | 53 (12) | 58 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 4 | 16
  Male | 2 | 2 | 2 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 5 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 2 | 7
  White | 4 | 3 | 3 | 3 | 13
  More than one race | 0 | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
GERD symptom severity [Mean (Standard Deviation); unit: scores on a scale] — GERD symptom severity was calculated by averaging the severity of GERD symptoms over a 7 day period based on the sum of scores from daily symptom diaries assessing the severity of daytime heartburn, nighttime heartburn, and acid reflux each on a 0-4 point scale (none, mild, moderate, severe, very severe). Higher scores signify worse symptoms (range 0-12).
  scores on a scale | 4.2 (2.1) | 5.6 (2.6) | 3.6 (2.2) | 3.8 (2.3) | 4.3 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Safety - Number of Participants Experiencing a Serious Adverse Event
Description: Serious adverse events (as defined by the FDA) are events that are potentially life-threatening or result in death, hospitalization, an emergency room visit, disability or permanent damage, a congenital abnormality, require intervention to prevent permanent impairment, or seriously jeopardizes a patient's health.
Time Frame: 2 week follow-up
Population: All enrolled study participants.
Measure: Number; unit: participants
Arm/Group | Placebo + Standard Interview | Supplement + Standard Interview | Placebo + Expanded Interview | Supplement + Expanded Interview
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Subjects With a 50% or Greater Decrease in GERD Symptom Severity
Description: Average daily GERD symptom severity during the last 7 days of the study was compared to average daily GERD symptom severity at baseline using daily study diary entries. GERD symptom severity for each day was based on the sum of scores assessing the severity of daytime heartburn, nighttime heartburn, and acid reflux each on a 0-4 point scale (none, mild, moderate, severe, very severe). Higher scores signify worse symptoms. The number of subjects with a 50% or greater decrease in GERD symptom severity from baseline to end of study in each group was calculated.
Time Frame: Second week of the trial compared to pre-trial baseline
Population: All enrolled study participants.
Measure: Number; unit: participants
Arm/Group | Placebo + Standard Interview | Supplement + Standard Interview | Placebo + Expanded Interview | Supplement + Expanded Interview
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants | 2 | 0 | 5 | 4
Statistical Analysis 1: Comparison: Placebo + Standard Interview vs Supplement + Standard Interview vs Placebo + Expanded Interview vs Supplement + Expanded Interview; All 4 arms were combined to compare the Standard Interview groups to the Expanded Interview groups. We calculated that we had 45-74% power to detect a 30-40% difference in responders between groups in the pre-specified primary outcome measure, the percent of subjects with a 50% or greater improvement in GERD symptom severity; Test type: Superiority or Other; p = 0.01, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo + Standard Interview vs Supplement + Standard Interview vs Placebo + Expanded Interview vs Supplement + Expanded Interview; All 4 arms were combined to compare the Placebo groups to the Supplement groups. We calculated that we had 45-74% power to detect a 30-40% difference in responders between groups in the pre-specified primary outcome measure, the percent of subjects with a 50% or greater improvement in GERD symptom severity; Test type: Superiority or Other; p = 0.33, Regression, Logistic

3. Secondary Outcome: GERD Health-Related Quality of Life at Follow-up
Description: The GERD Health-Related Quality of Life (GERD-HRQL) scale is a validated instrument assessing GERD-specific health-related quality of life using 10 questions, each on a 0-5 point scale. Scale range is 0-50 with higher numbers signifying worse quality of life.
Time Frame: Two weeks
Population: All enrolled study participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Standard Interview | Supplement + Standard Interview | Placebo + Expanded Interview | Supplement + Expanded Interview
Number analyzed (Participants) | 6 | 6 | 6 | 6
units on a scale | 18.2 (4.5) | 26.3 (7.8) | 17.7 (3.4) | 18.3 (4.9)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Data collected from subject symptom diaries.
Arm/Group | Placebo + Standard Interview | Supplement + Standard Interview | Placebo + Expanded Interview | Supplement + Expanded Interview
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 1/6 | 4/6 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Standard Interview (N=6) | Supplement + Standard Interview (N=6) | Placebo + Expanded Interview (N=6) | Supplement + Expanded Interview (N=6)
Cramping or abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 1 | 1 — Subject-reported symptom on daily symptom diary, may not be a true adverse event.
Diarrhea or loose stools (Gastrointestinal disorders) | 2 | 0 | 1 | 0 — Subject-reported symptom on daily symptom diary, may not be a true adverse event.
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 — Subject-reported symptom on daily symptom diary, may not be a true adverse event.
Heartburn (Gastrointestinal disorders) | 1 | 1 | 2 | 1 — Subject-reported symptom on daily symptom diary, may not be a true adverse event.
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 0 — Subject-reported symptom on daily symptom diary, may not be a true adverse event.
Burping (Gastrointestinal disorders) | 0 | 0 | 1 | 1 — Subject-reported symptom on daily symptom diary, may not be a true adverse event.
Headache (Nervous system disorders) | 2 | 0 | 0 | 2 — Subject-reported symptom on daily symptom diary, may not be a true adverse event.
Cough or congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Subject-reported symptom on daily symptom diary, may not be a true adverse event.
Nausea and/or vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0 — Subject-reported symptom on daily symptom diary, may not be a true adverse event.
Throat or mouth discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — Subject-reported symptom on daily symptom diary, may not be a true adverse event.
Sweating (General disorders) | 0 | 0 | 1 | 0 — Subject-reported symptom on daily symptom diary, may not be a true adverse event.
Fatigue (General disorders) | 1 | 0 | 0 | 1 — Subject-reported symptom on daily symptom diary, may not be a true adverse event.
Bright red blood per rectum (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — Subject-reported symptom on daily symptom diary, may not be a true adverse event.
Chest pain (Cardiac disorders) | 0 | 0 | 0 | 1 — Subject-reported symptom on daily symptom diary, may not be a true adverse event.
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 — Subject-reported symptom on daily symptom diary, may not be a true adverse event.
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 — Subject-reported symptom on daily symptom diary, may not be a true adverse event.

LIMITATIONS AND CAVEATS:
Small, pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No